CLINICAL TRIAL: NCT00936975
Title: A Phase 2, Multicenter Evaluation of 18F-Fluoride PET as a Pharmacodynamic Biomarker for Dasatinib, a Src Kinase Inhibitor, in Men With Castration-Resistant Prostate Cancer and Bone Metastases (BMS #180-279)
Brief Title: Fluorine F 18 Sodium Fluoride Positron Emission Tomography in Evaluating Response to Dasatinib in Patients With Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2010-01292; NCI-2010-01292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000647592; ACRIN 6687 (Other: ECOG-ACRIN Cancer Research Group); ACRIN-6687 (Other: CTEP); U01CA080098 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2014-12

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Malignant Neoplasm in the Bone; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- 18F-Fluoride PET (Experimental): Patients undergo fluorine F 18 sodium fluoride PET scan at baseline and then at 12 weeks after initiation of treatment with dasatinib. Dasatinib was administered under a concurrent protocol and was not considered part of the intervention on this protocol
  Interventions: Radiation: Fluorine F 18 Sodium Fluoride

INTERVENTIONS:
Radiation: Fluorine F 18 Sodium Fluoride — Undergo fluorine F 18 sodium fluoride PET scan
  Other Names: 18 F-NaF; F-18 NaF

SUMMARY:
This phase II trial is studying how well fluorine F 18 sodium fluoride positron emission tomography (PET) works in evaluating response to dasatinib in patients with prostate cancer and bone metastases. Diagnostic procedures, such as fluorine F 18 sodium fluoride PET, may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if changes in regional fluoride incorporation, measured by 18F-fluoride PET (SUV and Ki), occur in both castration-resistant prostate cancer bone metastases and normal bone as a response to treatment with dasatinib.

SECONDARY OBJECTIVES:

I. Determine if changes in 18F-fluoride transport (K1), an indicator of blood flow, and therefore, an indirect marker of angiogenesis, occur in both castration-resistant prostate cancer bone metastases and normal bone as a response to treatment with dasatinib.

OUTLINE: This is a multicenter study.

Patients undergo fluorine F 18 sodium fluoride PET scan at baseline and then at 12 weeks after initiation of treatment with dasatinib. PET parameters (SUV, Ki, and Kl) are also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Men 18 years or older with metastatic castration-resistant prostate cancer enrolling onto the Febbo clinical trial with dasatinib therapy (must meet all inclusion criteria for dasatinib treatment study and comply with requirements of that specific clinical trial)
* Histologic confirmation of original prostate cancer diagnosis
* Presence of at least one convincing bone metastasis as defined by bone scintigraphy, computed tomography (CT) scan (magnetic resonance imaging [MRI] if indicated), or plain X-ray
* Must currently have castrate testosterone levels (< 50 ng/dL) from orchiectomy or maintenance on a luteinizing hormone-releasing hormone (LHRH) agonist or LHRH antagonist

Exclusion Criteria:

* On the nilutamide-only arm (Arm A of the clinical therapeutic trial)

  * Note: However, if a patient crosses-over from nilutamide at the time of progression to add dasatinib therapy, he may be eligible for 18F-fluoride PET imaging protocol if he meets all inclusion criteria for this trial
* Any condition that would alter the patient's mental status, prohibiting the basic understanding and/or authorization of informed consent
* A serious underlying medical condition that would otherwise impair the patient's ability to receive treatment and imaging studies
* Expected lifespan of 12 weeks or less
* Extremely poor intravenous access, prohibiting the placement of a peripheral IV line for injection of radiotracer
* Initiation of bisphosphonate therapy less than 4 weeks from the first PET scan
* Radiation treatment to bone less than 4 weeks from first PET scan
* Radiopharmaceutical treatment to bone less than 4 weeks from first PET scan
* Treatment with granulocyte-macrophage colony stimulating factor (GM-CSF) or granulocyte CSF (G-CSF) within 4 weeks prior to first PET scan
* Inability to lie still for the imaging
* Weight > 300 lbs. (due to equipment specifications)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Yu, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall: Participants on the parent study ("Genomic Guided Therapy with Dasatinib or Nilutamide in Metastatic Castration-Resistant Prostate Cancer") receiving 100mg PO QD Dasatinib
Period: Overall Study
Arm/Group | Overall
Started | 18
Completed | 12
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 3
Not completed — Post-Tx scan uninterpretable | 2

BASELINE CHARACTERISTICS:
Population: 18 participants meeting the eligibility criteria were accrued to the trial and received the baseline PET scan
Groups:
- Overall: Participants receiving 100mg PO QD Dasatinib with F18 Sodium Fluoride PET scans at baseline
Arm/Group | Overall
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Changes in 18F-fluoride PET (SUV) - Tumor Bone
Description: Investigation of changes between baseline and 12 weeks in regional fluoride incorporation as measured by 18F-fluoride PET in tumor bone as measured by SUVmax
Time Frame: Baseline and 12 weeks
Population: Analysis population consists of 37 bone locations in 12 participants who were eligible for the study and had interpretable Pre- and Post-Treatment PET scans
Measure: Mean (Standard Deviation); unit: SUVmax
Units Other Than Participants: Bone sites
Groups:
- 18F-Fluoride PET: Patients undergo fluorine F 18 sodium fluoride PET scan at baseline and then at 12 weeks after initiation of treatment with dasatinib. Scans are done of normal bone and tumor bone at each time point
  fluorine F 18 sodium fluoride: Undergo fluorine F 18 sodium fluoride PET scan
Arm/Group | 18F-Fluoride PET
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
SUVmax | -6.67 (8.98)
Statistical Analysis 1: Comparison: 18F-Fluoride PET; This was an exploratory study and no a priori assumptions were employed; Test type: Superiority or Other; p < 0.001, GEE — GEEs were used to model the change in tumor uptake between baseline and 12 weeks. GEEs were used to adjust for the correlation of 37 tumors in 12 patients measured at 2 time points and to adjust for age as a confounder; Slope = -6.6084, Standard Error of Mean 1.7644 — GEEs, rather than a simple mean difference, were used to account for the multiple (clustered) bone measurement values within a patient and to adjust for age so that appropriate SE estimates (and thus p-values) were produced

2. Secondary Outcome: Changes in 18F-fluoride Transport (by Patlak Flux) - Tumor
Description: Investigation of changes in regional fluoride incorporation as measured by 18F-fluoride transport (Patlak flux) in Tumor. This measurement uses the Patlak method for determining the influx constant.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mL/min/mL
Units Other Than Participants: Bone sites
Groups:
- Overall: Participants receiving 100mg PO QD Dasatinib
Arm/Group | Overall
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
mL/min/mL | -0.01 (0.06)
Statistical Analysis 1: Comparison: Overall; the difference in Patlak flux in tumor bone between baseline and 12 weeks, accounting for the fact that each participant could contribute more than one tumor bone; Test type: Superiority or Other; p = 0.1945, GEE — [p-value comment as in outcome 1, analysis 1]; GEE was used to model the change, accounting for 37 tumors in 12 patients measured at 2 time points; Slope = -0.0115, Standard Error of Mean 0.0089 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Changes in 18F-fluoride PET SUV - Normal Bone
Description: Investigation of changes between baseline and 12 weeks in regional fluoride incorporation as measured by 18F-fluoride PET (SUV) in normal bone as measured by SUVmax
Time Frame: Baseline and 12 weeks
Population: Analysis population consists of 37 normal bone locations in 12 participants who were eligible for the study and had interpretable Pre- and Post-Treatment PET scans
Measure: Mean (Standard Deviation); unit: SUVmax
Units Other Than Participants: Bone sites
Arm/Group | 18F-Fluoride PET
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
SUVmax | 0.31 (1.17)
Statistical Analysis 1: Comparison: 18F-Fluoride PET; Test type: Superiority or Other; p = 0.32, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]; GEE was used to model the change, accounting for 37 tumors in 12 patients measured at 2 time points; Slope = 0.33, Standard Error of Mean 0.3274 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 18F-Fluoride PET; H0: No difference in uptake b/w normal & tumor bones; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; Age was included in the model as a confounder; Slope = 6.98, Standard Error of Mean 1.6943 — Estimated value is the slope of the Normal bone. Tumor Bone was used as reference category. GEEs, rather than a simple mean difference, were used to account for clustering and correlation of bone measurement values within a patient

4. Primary Outcome: Changes in 18F-fluoride Ki - Tumor Bone
Description: Investigation of changes between baseline and 12 weeks in regional fluoride incorporation as measured by 18F-fluoride PET (Ki) in tumor bone. Ki represents the net uptake of fluoride to the bone mineral compartment and reflects the level of osteoblastic activity in bone
Time Frame: Baseline and 12 weeks
Population: Analysis population consists of 37 Tumor bone locations in 12 participants who were eligible for the study and had interpretable Pre- and Post-Treatment PET scans
Measure: Mean (Standard Deviation); unit: mL/min/mL
Units Other Than Participants: Bone sites
Arm/Group | 18F-Fluoride PET
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
mL/min/mL | -0.02 (0.07)
Statistical Analysis 1: Comparison: 18F-Fluoride PET; Test type: Superiority or Other; p = 0.16, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; GEE was used to model the change, accounting for 37 tumors in 12 patients measured at 2 time points; Slope = -0.0177, Standard Error of Mean 0.0125 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Changes in 18F-fluoride Ki - Normal Bone
Description: Investigation of changes between baseline and 12 weeks in regional fluoride incorporation as measured by 18F-fluoride PET (Ki) in normal bone. Ki represents the net uptake of fluoride to the bone mineral compartment and reflects the level of osteoblastic activity in bone
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/mL
Units Other Than Participants: Bone sites
Arm/Group | 18F-Fluoride PET
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
mL/min/mL | 0.0 (0.01)
Statistical Analysis 1: Comparison: 18F-Fluoride PET; Test type: Superiority or Other; p = 0.53, Generalized Estimating Equation; GEE was used to model the change, accounting for 37 tumors in 12 patients measured at 2 time points; Slope = 0.0017, Standard Error of Mean 0.0027 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 18F-Fluoride PET; H0: influx(Ki) is the same in normal and tumor bones; Test type: Superiority or Other; p = 0.1095, Generalized estimating equations — [p-value comment as in outcome 1, analysis 1]; Age was included in the model as a confounder; Slope = 0.0205, Standard Error of Mean 0.0128 — [estimate comment as in outcome 3, analysis 2]

6. Secondary Outcome: Changes in 18F-fluoride Transport (by Patlak Flux) - Normal
Description: Investigation of changes in regional fluoride incorporation as measured by 18F-fluoride transport (Patlak flux) in normal bone. Palak flux is an indicator of blood flow and an indirect marker of angiogenesis.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mL/min/mL
Units Other Than Participants: Bone sites
Arm/Group | Overall
Number analyzed (Participants) | 12
Number analyzed (Bone sites) | 37
mL/min/mL | 0.01 (0.01)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.0033, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; GEE was used to model the change, accounting for 37 bones in 12 patients measured at 2 time points; Slope = 0.0061, Standard Error of Mean 0.0021 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Overall; H0: Change Patlak Flux from TP1 to TP2 is the same in normal and tumor bones; Test type: Superiority or Other; p = 0.0670, Generalized estimating equations — [p-value comment as in outcome 1, analysis 1]; Age was included in the model as a confounder; Slope = 0.0177, Standard Error of Mean 0.0097 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Overall; H0: %Change in Patlak Flux between timepoint 1 and 2 is the same for Normal and Tumor bones; Test type: Superiority or Other; p = 0.0278, Generalized estimating equations — [p-value comment as in outcome 1, analysis 1]; Slope = 32.3288, Standard Error of Mean 14.6956 — [estimate comment as in outcome 3, analysis 2]

ADVERSE EVENTS:
Time Frame: Only AEs that occur within 24 hours (± 4 hours [approximately 10 half lives]) of 18F-fluoride administration will be reported
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less